CLINICAL TRIAL: NCT03545438
Title: Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of LIB003 in Healthy Subjects With Hypercholesterolemia on Diet or Statin Therapy
Brief Title: Study to Evaluate the Safety, PK, and Pharmacodynamics of LIB003
Acronym: LIB003SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: LIB003-001
Record Dates: First submitted 2018-04-19; First posted 2018-06-04 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: single ascending dose with placebo controll
Who Masked: Participant, Care Provider, Investigator
Masking Description: Within each dosing cohort randomization is performed according to a computer-generated randomization scheme. Other than the study drug prepared by an unblinded pharmacist and administered by unblinded nurses who will be instructed not to discuss randomized treatment assignments and have no other role in the study, all study staff and PI, along with the subjects are blinded as to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- cohort 1 (Placebo Comparator): LIB003 dose 1 SC
  Interventions: Biological: LIB003
- cohort 2 (Placebo Comparator): LIB003 dose 2 SC
  Interventions: Biological: LIB003
- cohort 3 (Placebo Comparator): LIB003 dose 4 SC
  Interventions: Biological: LIB003
- cohort 4 (Placebo Comparator): LIB003 dose 4 SC
  Interventions: Biological: LIB003
- cohort 5 (Placebo Comparator): LIB003 dose 5 SC
  Interventions: Biological: LIB003
- cohort 6 (Placebo Comparator): LIB003 dose 4 IV
  Interventions: Biological: LIB003
- cohort 7 (Placebo Comparator): LIB003 dose 5 IV
  Interventions: Biological: LIB003
- cohort 8 (Placebo Comparator): LIB003 dose 3 SC - statin treated
  Interventions: Biological: LIB003
- cohort 9 (Placebo Comparator): LIB003 dose 4 SC - statin treated
  Interventions: Biological: LIB003

INTERVENTIONS:
Biological: LIB003 — LIB003 or placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, single ascending dose study in nine (9) separate and sequential dose cohorts (7 SC and 2 IV cohorts) to assess the safety and tolerability, pharmacokinetics and pharmacodynamics of LIB003 in subjects with moderately elevated LDL-C levels.

DETAILED DESCRIPTION:
After meeting eligibility criteria within each cohort subjects will be randomized to receive a single dose of LIB003. Seven (7) cohorts will receive LIB003 escalating doses of LIB003, or placebo, by SC injection and 2 cohorts LIB003 or placebo by IV infusion. Dose escalation will be based on the assessment of safety and tolerability data. All cohorts will each first enroll a sentinel group of subjects who will receive LIB003 or placebo in a double-blind fashion with the remaining subjects in that cohort only to be dosed after the safety data on day 4 from the sentinel subjects has been assessed and deemed safe.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are >/=18 and </=70 years of age. Female subjects must be of non-childbearing potential.
* LDL-C >/=100 mg/dL who are either not on a lipid-lowering therapy or who are on stable statin therapy.
* Body mass index (BMI) >18 and <38 kg/m2
* Mild hypertensives on a stable dose of no more than one antihypertensive drug

Exclusion Criteria:

* History of any prior or concomitant clinical condition or acute and/or unstable systemic disease compromising subject inclusion
* Systolic blood pressure <90 mmHg or >160 mmHg or diastolic blood pressure <50 or >100 mmHg at screening
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C virus antibody
* Abnormal liver function test at Screening (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >2 × the upper limit of normal [ULN]
* Estimated glomerular filtration rate <60 mL/min/1.73 m2 at screening, as determined by the CKD-EPI Equation
* History of prescription drug abuse, illicit drug use (including marijuana), or alcohol abuse
* Unable to spend 4 days in confinement unit
* History of allergy to protein-based biologics including, but not limited to, mAbs and vaccine
* Any other finding which, in the opinion of the Investigator, would compromise the subject's safety or participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of treatment emergent adverse events (TEAEs) | 43 days
  safety and tolerability will be assessed by the incidence and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
Absolute change in serum unbound (free) proprotein convertase subtilisin/kexin type 9 (PCSK9) concentrations over time | 43 days
  Serum free PCSK9 will be measured at baseline and various time points over 43 days
Absolute change in serum total PCSK9 over time | 43 days
  Serum total PCSK9 will be measured at baseline and various time points over 43 days
Percent change in Low Density Lipoprotein cholesterol (LDL-C) over time | 43 days
  Serum LDL-C will be measured at baseline and various time points over 43 days to derive percent change
Percent change in Apolipoprotein B (Apo B) over time | 43 days
  Serum Apo B will be measured at baseline and various time points over 43 days to derive percent change
Changes in serum LIB003 concentrations over time | 43 days
  serum LIB003 will be measured at various time points to derive AUC (area under curve)
Presence of anti LIB003 antibodies (ADAs) | 43 days
  Measurement of ADAs will be done at baseline and various intervals after LIB003 administration

CONTACTS AND LOCATIONS:
Overall Officials: Traci A Turner, MD, Principal Investigator — Medpace Clinical Research
Locations (1):
- Medpace (MARC/CPU), Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-11-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03545438/Prot_000.pdf